CLINICAL TRIAL: NCT01740453
Title: Interscalene Block on Ventilatory Function After Shoulder Surgery : Evaluation of Single or Continuous Injection
Brief Title: Effect of Interscalene Block on Ventilatory Function
Acronym: KTBIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, MD, PhD, Centre Hospitalier Universitaire de Nīmes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTBIS-2012-V1
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Respiratory Depression; Anesthesia Morbidity; Block
MeSH Terms: conditions — Respiratory Insufficiency; Bites and Stings | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single (no catheter) (No Intervention): ropivacaine single injection : 5 mg/ml 15 ml
- Continuous infusion (Experimental): Single injection with continuous injection ropivacaine 2 mg/ml 8 ml/h
  Interventions: Drug: ropivacaine 2 mg/ml

INTERVENTIONS:
Drug: ropivacaine 2 mg/ml — single
  Arms: Continuous infusion

SUMMARY:
Interscalene block with local anesthetic impairs ventilation (unilateral diaphragmatic dysfunction). Single injection of local anesthetic induced transitory dysfunction (< 24h). The investigators hypothesized that continuous interscalene block would prolonged ventilatory impairment

DETAILED DESCRIPTION:
Unilateral pulmonary dysfunction occured after interscalene block due to phrenic nerve paralysis. This reduction induced vital capacity alteration and peek flow reduction.Several studies analysed dysfunction recovery duration after single injection using short (lidocaine)or intermediate (ropivacaine, bupivacaine)local anesthetic drug. Because continuous infusion prolonged block duration, phenic nerve may be also prolonged. However no study with continuous interscalene infusion have been performed for this dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* surgery : scheduled for elective shoulder surgery
* available for 1 month of follow up
* physical status : 1, 2, 3

Exclusion Criteria:

* body mass index > 35
* contraindication for interscalene block (local sepsis, bleeding, allergy, peripheral neuropathy)
* vital capacity less than 1.5 liters
* cardiac or renal insufficiency
* physical status >3, pregnant, weigh less than 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction of the pulmonary forced vital capacity | Day 2
  A 25 % reduction of the pulmonary forced vital capacity is expected and measured using spirometer

SECONDARY OUTCOMES:
Reduction of the pulmonary maximum forced expiratory flow | Day 2
  Outcome measure was performed using a spirometer
Morphine consumption | Day 2
  Additional morphine administration for pain management (morphine intravenous : 1 mg every 7 min when necessary, pain score > 3/10)
Pain score at rest and motion | Day 2
  Outcome Measure using a visual analog scale (0 to 10)

OTHER OUTCOMES:
Duration of sensory interscalene block | Day 2
  outcome measure was performed using a cold test on the skin

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cuvillon, Md,PhD, Principal Investigator — Caremeau Hospital, Nimes, France
Locations (1):
- Centre hospitalier La Pitié Salpetriere, Paris, Île-de-France Region, France